CLINICAL TRIAL: NCT03911505
Title: An Open-label Study of the Safety, Pharmacokinetics, Efficacy, Pharmacodynamics, and Immunogenicity of Cipaglucosidase Alfa/Miglustat in Pediatric Subjects Aged 0 to < 18 Years With Late-onset Pompe Disease
Brief Title: ZIP Study-OL Study of Safety, PK, Efficacy, PD, Immunogenicity of ATB200/AT2221 in Pediatrics Aged 0 to < 18 y.o. w/LOPD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATB200-04
Expanded Access: NCT03865836 (Available)
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Pompe Disease (Late-onset)
Keywords: Pompe; rhGAA
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — miglustat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cipaglucosidase Alfa (ATB200)/Miglustat(AT2221) (Experimental): Participants received Cipaglucosidase Alfa (ATB200) co-administered with Miglustat (AT2221) capsule
  Interventions: Biological: Cipaglucosidase Alfa; Drug: Miglustat

INTERVENTIONS:
Biological: Cipaglucosidase Alfa — Enzyme Replacement Therapy via intravenous infusion
  Other Names: ATB200
Drug: Miglustat — Participants received Cipaglucosidase Alfa (ATB200) co-administered with Miglustat(AT2221)
  Other Names: AT2221

SUMMARY:
This is a Phase 3, open-label, multicenter study to evaluate the safety, PK, efficacy, PD, and immunogenicity of Cipaglucosidase Alfa/Miglustat treatment in enzyme replacement therapy (ERT)-experienced and ERT-naïve pediatric subjects with Pompe disease, aged 0 to < 18 years

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects (ERT-naïve [have never received a dose of rhGAA] or ERT-experienced [have received rhGAA every 2 weeks for at least 6 months immediately before enrollment, and if ERT dosage has been modified, must have been on the modified dosage for at least 3 months before enrollment]) diagnosed with LOPD who are aged 12 to <18 years at screening (Cohort 1 only) or aged 0 months to < 12 years at screening (Cohort 2 only)
2. Subject weighs ≤ 115 kg. (Cohort 1 Only)
3. Subject must have a diagnosis of LOPD based on documentation as defined in study protocol
4. If of reproductive potential and if sexually active, female and male subjects agree to use a highly effective method of contraception throughout the duration of the study and for up to 90 days after their last dose of Cipaglucosidase Alfa/Miglustat
5. Subject has a sitting forced vital capacity (FVC) ≥ 30% of the predicted value for healthy Adolescents at screening (Cohort 1 only)
6. Subject (aged 12 to <18 years; Cohort 1) performs one 6-Minute Walk Test (6MWT) (≥ 75 meters) at screening that is valid, as determined by the clinical evaluator, or subject (aged ≥ 5 to < 12 years; Cohort 2) performs one 6MWT (≥ 40 meters) at screening that is valid, as determined by the clinical evaluator

Exclusion Criteria:

1. Subject has received any investigational/experimental drug, oral anabolic steroid or derivative, biologic, or device within 30 days or 5 half-lives of the therapy or treatment, whichever is longer, before screening
2. Subject has received treatment with prohibited medications within 30 days of screening
3. Subject has received any gene therapy at any time
4. Subject has any intercurrent illness or condition at screening or baseline that may preclude the subject from fulfilling the protocol requirements or suggests to the investigator and/or the medical monitor that the potential subject may have an unacceptable risk by participating in this study
5. Subject has a hypersensitivity to any of the excipients in ATB200, approved rhGAA, or AT2221
6. Female subject is pregnant or breast-feeding at screening
7. Subject requires the use of ventilation support for > 6 hours per day while awake
8. Subject has evidence of moderate to severe hypertrophic cardiomyopathy aligning with classic IOPD
9. In the opinion of the investigator, the parent or legally authorized representative is unlikely or unable to comply with the study requirements
10. Subject has any prior history of illness or condition known to affect motor function, such as, but not limited to, Guillain-Barre syndrome, cerebral palsy, etc
11. Subject who is diagnosed with Pompe disease via newborn screening and is asymptomatic (ie, showing no signs and symptoms of Pompe disease (Cohort 2 Only)

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) from baseline | 52 weeks

SECONDARY OUTCOMES:
Assessment of pharmacokinetic parameters | 52 weeks
  ATB200 and AT2221 concentrations in plasma

CONTACTS AND LOCATIONS:
Locations (17):
- United States (9):
  - University of Florida Clinical Research Center, Gainesville, Florida
  - Wolfson Children's Hospital, Jacksonville, Florida
  - Woodruff Memorial Research Building, Atlanta, Georgia
  - St. Louis Children's Hospital, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Clinical and Translational Sciences Institute, Salt Lake City, Utah
  - Lysosomal and Rare Disorders Research and Treatment Center, Inc., Fairfax, Virginia
- Women's and Children's Hospital, North Adelaide, South Australia, Australia
- University of Calgary, Calgary, Alberta, Canada
- SphinCS GmbH Clinical Science for LSD, Hochheim am Main, Hesse, Germany
- San Gerardo Hospital, Monza, Italy
- Japan (4):
  - Izumi City General Hospital, Osaka, Izumi-Shi
  - Gunma University Hospital, Gunma
  - Tohoku University Hospital, Miyagi
  - Tokyo Women's Medical University, Tokyo

IPD SHARING:
Plan to Share IPD: No